CLINICAL TRIAL: NCT01944982
Title: Salvage Therapy With Chemotherapy and Natural Killer Cells in Relapsed/Refractory Paediatric T Cell Lymphoblastic Leukaemia and Lymphoma.
Acronym: HNJ-NKAES-2012
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The low recruitment rate makes it very difficult to complete the study within a reasonable period of time.
Sponsor: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Responsible Party: Principal Investigator, Antonio Perez-Martinez, Doctor, Hospital Universitario La Paz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNJ-NKAES-2012; 2012-000054-63 (EudraCT Number)
Record Dates: First submitted 2013-09-13; First posted 2013-09-18 (Estimated); Last update posted 2016-12-20 (Estimated); Status verified 2016-12

CONDITIONS: Relapsed/Refractory Paediatric T Cell Lymphoblastic Leukaemia and Lymphoma
Keywords: Immunotherapy; NKAEs; Expanded haploidentical natural killer cells; Activated natural killer cells
MeSH Terms: conditions — Recurrence; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Activated natural killer cells (Experimental): Activated natural killer cells
  Interventions: Biological: Expanded haploidentical natural killer cells (NKAEs)

INTERVENTIONS:
Biological: Expanded haploidentical natural killer cells (NKAEs)

SUMMARY:
To determine safety profile of immunotherapy with natural killer cells and activated expanded (NKAEs) after salvage chemotherapy in relapsed/refractory paediatric T cell lymphoblastic leukaemia and lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 0 and 21 years with relapsed or refractary acute lymphoblastic leukemia or T-cell lymphoblastic lymphoma.
* Lansky Index > 60%.
* Left ventricular ejection fraction > 39%.
* Negative HIV serology.
* Provide informed consent in accordance with current legislation.

Exclusion Criteria:

* Patients with a history of poor compliance.
* Patients not valid after psycho-social evaluation
* Severe (4) functional organ disorders (hepatic, renal, respiratory) according to NCI CTCAE v3 criteria

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2013-07; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Safety profile (number of AEs per patient) | Two months

SECONDARY OUTCOMES:
Incidence of episodes of febrile neutropenia, bacteriemia or viral or fungal infections | During 14 months
time to hematological recovery (days) | 2 months
  hematological recovery: neutrophils >500/mm3, lymphocytes >250/mm3 and platelets >50.000/mm3)
days of hospitalization in each cycle | 2 months
Objective response rate | 2 months
  Objective response rate according to cytomorphic and by "minimal residual disease" criteria (cytometry and/or real time PCR)
days of isolation | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pérez-Martínez, MD, PhD, Principal Investigator — Service of Pediatric Hematology-Oncology
Locations (1):
- Pediatric Hematology-Oncology; Hospital Infantil Universitario La Paz, Madrid, Madrid, Spain

REFERENCES:
- [Derived] Vela M, Corral D, Carrasco P, Fernandez L, Valentin J, Gonzalez B, Escudero A, Balas A, de Paz R, Torres J, Leivas A, Martinez-Lopez J, Perez-Martinez A. Haploidentical IL-15/41BBL activated and expanded natural killer cell infusion therapy after salvage chemotherapy in children with relapsed and refractory leukemia. Cancer Lett. 2018 May 28;422:107-117. doi: 10.1016/j.canlet.2018.02.033. Epub 2018 Feb 23. PMID 29477379